CLINICAL TRIAL: NCT06358378
Title: Accuracy of Cuffless Ambulatory Blood Pressure Monitors Compared to Cuff-based Monitors in an Ambulatory Elderly Population: A Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sligo General Hospital (Other)
Responsible Party: Principal Investigator, Zaran Butt, Cardiology Specialist Registrar, Sligo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 995
Record Dates: First submitted 2024-03-31; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Enrolled patients will be asked to wear both the cuff-based ambulatory blood pressure monitor (ABPM) and the Aktiia bracelet at the same time during daytime hours (9am - 9pm) for a 72-hour period after calibration of the bracelet at the site. The ABPM will provide reference blood pressure measures to compare the Aktiia-derived measures against
  Interventions: Device: Aktiia SA Bracelet

INTERVENTIONS:
Device: Aktiia SA Bracelet — The Aktiia device is a wearable blood pressure monitor developed by the company Aktiia SA. It is designed to monitor at blood pressure frequent intervals throughout the day and night without the need for inflatable cuffs. Instead, it contains optical sensors which collect photoplethysmography signals from arteries in the patient's wrist and uses these to estimate blood pressure. The device only takes measurements when it perceived optimal conditions for doing so, corresponding to minimal arm movement (i.e. a resting state) for at least five minutes and good quality signal detection. This device is commercially available and validated for use in adults aged 85 and younger.

SUMMARY:
Hypertension is extremely common amongst the elderly, typically manifesting as a silent disease with potentially devastating consequences if left undetected and untreated. Such consequences include stroke, myocardial infarction, kidney and eye disease. Opportunistic screening for hypertension is therefore standard in clinical practice. Currently, the standard of care for screening in the western world is with 24-hour ambulatory cuff-based devices which are often intolerable, particularly for elderly patients.

Several novel cuffless wearables have been developed to overcome the limitations of cuff-based monitors. These devices offer significant advantages over cuff-based devices, including improved patient tolerance and user acceptability. Numerous cuffless monitors are now commercially available. However, validation of such devices is challenging as there is no current universal standard for validating such devices.5 This is highlighted by the heterogenous and often inadequate study methods used to demonstrate accuracy of commercially available cuffless devices for blood pressure measurements. Indeed, the uncertainty about their merit is reflected in international guidelines. The 2023 European Society of Hypertension guidelines currently do not recommend routine use of such devices in clinical practice for evaluation of blood pressure.

There are limited clinical trials comparing 24-hour cuff-based devices directly to cuffless devices, and even fewer specifically in an elderly population where they may be particularly advantageous due to design features that improve tolerability. This study thus aims to address this important gap in the literature to better understand if cuffless devices provide reliable blood pressure measurements in the elderly population by directly comparing these devices to the current standard of care in blood pressure evaluation. The Aktiia device will be used as a surrogate for cuffless wearables while a standard 24-hour ambulatory cuff-based device will represent cuff-based devices. The Aktiia device is a cuffless solution worn as a bracelet on the wrist. It contains optical sensors which collect photoplethysmography signals from arteries in the patient's wrist and uses these to estimate blood pressure. This device is commercially available and clinically validated for use in patients up to age 85.

ELIGIBILITY:
Inclusion Criteria:

* Adults >65 years old
* Enrolled on Sligo/Leitrim ICPOP programme
* Participants (or carers) must have access to a smart phone compatible with the Aktiia app

Exclusion Criteria:

* Cognitive impairment or diagnosis of dementia
* Adults unable to provide informed consent
* Life-expectancy less than one year
* Patient's unlikely to comply with trial protocol in opinion of investigator's

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean paired difference between cuffless daytime blood pressure measurements (systolic and diastolic) and cuff-based measurements | 4 months

SECONDARY OUTCOMES:
Mean paired difference between cuffless daytime blood pressure measurements (systolic and diastolic) and cuff-based measurements taken in a resting state | 4 months
Mean difference between mean 24-hour cuffless daytime blood pressure measurements (systolic and diastolic) and cuff-based measurements on a per patient basis | 4 months
Tolerability : Mean paired differences on Comfort Rating Scale (CRS) between devices | 4 months
  This is a well-validated, quick and easy-to-use tool to compare comfort of wearable devices.7 It consists of 6 domains of comfort, with a 21-point scale used to score each. A score of 0 indicates a high-level of comfort for a particular domain description, and vice versa for a score of 20. The mean and standard deviation will be reported for all domains, and compared across the two devices.
User Acceptability: Mean paired differences on System Usability Scale (SUS) between devices | 4 months
  This is a widely used, quick and well-validated questionnaire for the assessment of perceived usability. It consists of 10 items represented as statements relating to an aspect of usability. Each item is scored from 0-5 on a Likert scale, where '0' correlates to strong disagreement and '5' correlates to strong agreement. Overall transformed score ranges from 0 - 100, with higher scores indicating better user acceptability.

OTHER OUTCOMES:
Proportion of recruited patients who provide at least 5 daytime cuffless blood pressure readings per day | 4 months
  Pilot Outcome
Proportion of total measurements taken which can be paired (i.e. taken within 1-hour of a measurement from the other device) | 4 months
  Pilot Outcome
Proportion of missing data from activity diaries | 4 months
  Pilot Outcome
Proportion of recruited patients who provide at least 3 paired blood pressure readings for 3 consecutive days | 4 months
  Pilot Outcome

IPD SHARING:
Plan to Share IPD: Undecided